CLINICAL TRIAL: NCT04676074
Title: Effect of Upper Limb Ergometer on the Arthrogenic Index of Plasma in Post Menopausal Obese Women.
Brief Title: Effect of Upper Limb Ergometer on the AIP in Post Menopausal Obese Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Elbanna, lecturer at faculty of physical therapy at Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rana Hesham
Record Dates: First submitted 2020-12-11; First posted 2020-12-19 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Post Menopausal Obese Women

STUDY DESIGN:
Intervention Model Description: Participants had randomly divided into two equal groups. Group (A) which is the control group receive normal routine medication. Group (B) will receive normal routine medication with the treatment program of moderate intensity upper limb ergometer for 15 minute with frequency three times per week for four weeks.
Who Masked: Participant
Masking Description: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): the participant will not do any exercise program but just they will take the routine medication.
- study group (Experimental): will receive normal routine medication with the treatment program of moderate intensity upper limb ergometer for 15 minute with frequency three times per week for four weeks.
  Interventions: Device: Electronic Upper limb( body) ergometer

INTERVENTIONS:
Device: Electronic Upper limb( body) ergometer — Electronic pedal for the upper limb using for training the upper body. Intensity, speed and resistance can be adjusted.
  Arms: study group

SUMMARY:
Participants had randomly divided into two equal groups. Group (A) which is the control group receive normal routine medication. Group (B) will receive normal routine medication with the treatment program of moderate intensity upper limb ergometer for 15 minute with frequency three times per week for four weeks.

DETAILED DESCRIPTION:
Control group (A):

1. Each participant will sign a consent form after receiving a detailed explanation about the procedure.
2. A blood sample will been taken by a nurse in a heparinized tube and delivered to lab within six hours.
3. BMI will been measured body weight(Kg) and height (m2)

   a. BMI= body weight (Kg)/ height (m2).
4. Waist circumference will be measured.
5. After one month blood analysis evaluation will be done to record the response to the routine medication.

Training Procedure for group (B):

1. Each participant will sign a consent form after receiving a detailed explanation about the procedure.
2. A blood sample will been taken by a nurse in a heparinized tube and delivered to lab within six hours.
3. BMI will been measured body weight(Kg) and height (m2)

   a. BMI= body weight (Kg)/ height (m2).
4. Waist circumference will be measured.
5. The maximum heart rate will be determined from Tanaka formula (208- 0.7 *age of the participant)

   * Then the exercise load will be determined according heart rate reserve of the participants ( maximum heart rate - resting heart rate).
6. Start with sitting resting without any effort for 5 min then Start at a low speed and intensity for 5 minutes to warm up the body.
7. Increase the speed and intensity for 10-30 seconds before dropping it back for 2-5 minutes and Repeat according to the intensity.
8. Finally, a five minutes of cooling down with no resistance had performed.
9. After one month blood analysis evaluation will be done to record the response to the routine medication.

ELIGIBILITY:
Inclusion Criteria:

* female aged 45-60 years old.
* class 1 and 2 obesity.
* post menopausal.
* diagnosed as controlled diabetic.
* diagnosed as controlled hypertensive.

Exclusion Criteria:

* uncontrolled diabetic.
* uncontrolled hypertensive.
* class 3 and morbid obesity.
* mentally unstable person.
* Any shoulder, hand and elbow orthopedic or neural disorders.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Post Menopausal Obese Women
Enrollment: 40 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Effect of the upper body ergometer on arthrogenic index ( triglyceride/ high density lipoprotein) | after one month of the trial application
  Effect of the upper body ergometer on arthrogenic index ( triglyceride/ high density lipoprotein)

SECONDARY OUTCOMES:
Effect of the upper body ergometer on total body weight kg. | after one month of the trial application
  Effect of the upper body ergometer on total body weight kg.
Effect of the upper body ergometer on estimated maximum heart rate(beat/min). | after one month of the trial application
  Effect of the upper body ergometer on estimated maximum heart rate(beat/min).

CONTACTS AND LOCATIONS:
Overall Officials: Rana H El Banna, PHD, Principal Investigator — Faculty of physical therapy at Cairo University
Locations (1):
- Outpatient clinic faculty of physical therapy at Cairo University, Giza, Egypt